## **Informed Consent**

Effective Ads for Quitting Smoking

NCT06485479

06/20/2024

# University of North Carolina at Chapel Hill Consent to Participate in a Research Study

Consent Form Version Date: 6/20/2024

IRB Study # 23-2450

Title of Study: Communication about smoking study

**Principal Investigator:** Noel Brewer

Principal Investigator Department: Health Behavior Principal Investigator Email Address: ntb@unc.edu

Funding Source and/or Sponsor: National Institutes of Health (NIH)

#### **CONCISE SUMMARY.**

The purpose of this research study is to better understand people's cigarette use and their thoughts about a quit smoking campaign. The information we learn will help us ensure our campaign ads meet community members needs. Participants in this study will be asked to complete a short (15 minutes) online survey. Risks of being in the study are no greater than everyday life. There are no direct benefits to study participants. If you want to learn more about this study, please continue to read below.

## These are some things we want you to know about research studies:

You are being asked to take part in a research study. To join the study is voluntary. You may choose not to participate, or you may withdraw your consent to be in the study, for any reason, without penalty. Details about this study are discussed below. It is important that you understand this information so that you can make an informed choice about being in this research study.

#### Why are they doing this research study?

This study will examine a quit smoking campaign. The information we learn from this research will help us ensure our campaign ads meet community members needs.

## How many people will take part in this study?

There will be about 2,000 people in this research study.

#### What will happen during this study

You will complete an online survey where we ask you to view campaign ads designed to support people in quitting smoking. We will assign you to a study group by chance, like flipping a coin. After viewing the ads, participants will be asked to respond to survey items rating the ads. The survey will also ask items about health messages, tobacco laws, tobacco use, and demographics. The survey will last about 15 minutes.

#### Who will be told the things we learn about you in this study?

We will not tell anyone what you tell us without your permission unless there is something that could be dangerous to you or someone else. We will not ask for your name or any other identifying information from you in this study. Participants in this study *will not* be identified in any report or publication about this study. We may use de-identified data from this study in future research without additional consent.

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. With this Certificate, the researchers cannot be forced to disclose information that may identify you, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify you, except as explained below. The Certificate cannot be used to resist a demand for information from personnel of the United States Government that is

used for auditing or evaluation of Federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information.

#### What are the possible benefits from being in this study?

Research is designed to benefit society by gaining new knowledge. There are no direct benefits from being in this research study.

## What are the possible risks or discomforts involved from being in this study?

Risks of being in the study are no greater than everyday life. There may be uncommon or previously unknown risks. The only known risk of harm could come from a breach of confidentiality. There are no other known risks for this study. You should report any problems to the researcher.

## Will you receive anything for being in this study?

In the email you received that invited you to participate in the study, you were advised about your compensation amount from NORC. If you are unaware of this compensation amount, please review the invitation email.

#### Who should you ask if you have any questions?

For technical issues about the survey or questions about your compensation, please contact AmeriSpeak Support at <a href="mailto:support@AmeriSpeak.org">support@AmeriSpeak.org</a> or call (888) 326-9424. If you have other questions, complaints or concerns about your rights while you are in this research study you may contact the Institutional Review Board at 919-966-3113 or by email to IRB\_subjects@unc.edu.

| Participant's agreement: |
|---|
| I have read the information provided above. I have asked all the questions I have at this time. |
| I want to participate (survey starts) |
| I do NOT want to participate. (study ends) |